CLINICAL TRIAL: NCT01615705
Title: The Etiologic Role of Inflammation, Thrombophilia and Fibrinolysis in the Post-thrombotic Syndrome: The Bio-SOX Sub Study
Brief Title: Biomarker Sub Study of the Compression Stockings to Prevent the Post-Thrombotic Syndrome (SOX) Trial
Acronym: Bio-SOX
Status: Completed | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Sigvaris Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Susan Kahn, SOX Trial Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: MOP-89349/NA-5629; ISRCTN71334751 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-06-01; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Deep Venous Thrombosis
Keywords: Postphlebitic Syndrome; Post-Thrombotic Syndrome; Biomarkers; Markers of Inflammation; Genetic Thrombophilia; Coagulation Activation
MeSH Terms: conditions — Venous Thrombosis; Postphlebitic Syndrome; Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected and processed by centrifuge to obtain serum, peripheral blood leukocytes and platelet-poor plasma. Samples then aliquoted into 2.0ml microcentrifuge tubes for storage at -80°C until further analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood Draw: SOX Subjects:
  The cohort consists of original subjects from the SOX Trial who consented to participate in the sub study.

SUMMARY:
The purpose of this study is to evaluate whether biomarkers of inflammation, genetic thrombophilia and coagulation activation influence Post-Thrombotic Syndrome development in patients with symptomatic proximal deep venous thrombosis.

DETAILED DESCRIPTION:
The post-thrombotic syndrome (PTS) is a frequent, burdensome and costly condition that occurs in about one third of patients after an episode of deep vein thrombosis (DVT). Affected patients have chronic leg pain and swelling, and sometimes develop skin ulcers. Poor understanding of the pathophysiology and predictors of PTS has hampered progress in its prevention and treatment. Biomarkers reflective of inflammation, genetic thrombophilia and coagulation activation may be of value in predicting PTS development in patients with DVT; they may also provide insight into understanding the underlying mechanisms of PTS, which could result in the development and testing of novel therapies to prevent and treat PTS.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a first, symptomatic, objectively confirmed proximal DVT diagnosed within the last 14 days (with or without concurrent distal DVT or pulmonary embolism)
* Who have no contraindications to standard treatment with heparin and/or warfarin, and
* Who provide informed consent to participate

Exclusion Criteria:

* Contraindication to compression stockings Limited lifespan (estimated < 6 months)
* Geographic inaccessibility preventing return for follow-up visits
* Inability to apply stockings daily and unavailability of a caregiver to apply stockings daily
* Treatment of acute DVT with thrombolytic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously enrolled in the SOX Trial (ClinicalTrials.gov Identifier NCT00143598)
Sampling Method: Non-Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2004-06; Primary Completion 2010-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Markers of Inflammation | Baseline
  Blood samples drawn at baseline, 1 and 6-mths to evaluate the relationship between CRP, ICAM, IL-6, IL-10 with the subsequent development of PTS.
Markers of Inflammation | 1-mth follow up
  Blood samples drawn at baseline, 1 and 6-mths to evaluate the relationship between CRP, ICAM, IL-6, IL-10 with the subsequent development of PTS.
Markers of Other Thrombophilia | 6-mth follow up
  Blood samples drawn at 6-mths to evaluate the relationship between D-Dimer, VIII, Lupus anticoagulant, IgG, IgM with the subsequent development of PTS.
Markers of Inflammation | 6-month follow up
  Blood samples drawn at baseline, 1 and 6-mths to evaluate the relationship between CRP, ICAM, IL-6, IL-10 with the subsequent development of PTS.
Markers of Other Thrombophilia | 6-month follow up
  Blood samples drawn at 6-mths to evaluate the relationship between D-Dimer, VIII, Lupus anticoagulant, IgG, IgM with the subsequent development of PTS.

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Kahn, M.D., M.Sc., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (25):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
- Canada (22):
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences - Chedoke Division, Hamilton, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences - Henderson General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier Pierre-Boucher, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Sir Mortimer B. Davis -Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Hôpital Hôtel-Dieu, Montreal, Quebec
  - Royal Victoria Hospital - McGill University Health Centre, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec, Hôpital de l'Enfant-Jésus, Québec, Quebec

REFERENCES:
- [Background] Kahn SR, Shbaklo H, Shapiro S, Wells PS, Kovacs MJ, Rodger MA, Anderson DR, Ginsberg JS, Johri M, Tagalakis V; SOX Trial Investigators. Effectiveness of compression stockings to prevent the post-thrombotic syndrome (the SOX Trial and Bio-SOX biomarker substudy): a randomized controlled trial. BMC Cardiovasc Disord. 2007 Jul 24;7:21. doi: 10.1186/1471-2261-7-21. PMID 17711595
- [Derived] Rabinovich A, Cohen JM, Cushman M, Kahn SR; BioSOX Investigators. Association between inflammation biomarkers, anatomic extent of deep venous thrombosis, and venous symptoms after deep venous thrombosis. J Vasc Surg Venous Lymphat Disord. 2015 Oct;3(4):347-353.e1. doi: 10.1016/j.jvsv.2015.04.005. Epub 2015 Aug 1. PMID 26992609